CLINICAL TRIAL: NCT02397512
Title: Elucidating the Influence of Lactulose Intake on the Gut Microbiota Composition
Acronym: Lactulose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology in Zurich (ETHZ) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KEK-ZH-2014-0358
Record Dates: First submitted 2015-03-18; First posted 2015-03-25 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Changes in Gut Microbiota Composition After Lactulose Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulose group (Experimental): Subjects will ingest 50g of lactulose once
  Interventions: Drug: application of lactulose
- Control group (Placebo Comparator): Subjects will ingest 50g of sucrose once
  Interventions: Other: application of sucrose

INTERVENTIONS:
Drug: application of lactulose — Subjects will ingest 50g of lactulose once
  Arms: Lactulose group
Other: application of sucrose — Subjects will ingest 50g of sucrose once
  Arms: Control group

SUMMARY:
This study will test the influence of lactulose of the human gut microbiota. Healthy volunteers will ingest 50g of lactulose and donate stool samples 1 day before as well as 1-2 days and 14 days after the test. Using sequencing and metabolomics techniques the investigators will identify changes in microbiota composition upon lactulose exposure.

DETAILED DESCRIPTION:
This is a clinical study for investigating the influence of lactulose on the composition and metabolic activities of the intestinal microbiota. We will recruit 40 healthy volunteers. Subjects will be randomized and receive either 50g lactose (intervention group) or 50g sucrose (control group).

Subjects will donate fecal samples 24h before and after (1-2d, 14d) lactulose ingestion. After ingestion H2-in expiratory air and symptoms will be followed for 3 hours.

Frozen samples will be analyzed for their microbiota composition and key metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Subjects free of relevant abdominal complaints (=healthy)
* Written informed consent
* Working at ETH Zurich/University of Zurich, experience in handling of -80°C freezers on biosafety level 2

Exclusion Criteria:

* Previous history of gastrointestinal disease or surgery (excludes appendectomy, hernia repair and anorectal disorders)
* Known diabetes mellitus, scleroderma, neurological impairment or other major current disease
* Subjects unable to stop medication that alters gut flora: proton pump inhibitors, laxatives and antibiotics at least 4 weeks before study entry.
* Pregnancy beyond week 12 (no pregnancy test will be performed)
* Involvement in any other clinical trial during the course of this trial, nor within a period of 14 days prior to its beginning or 14 days after its completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Influence of lactulose intake on gut microbiota composition (microbiota sequencing, analysis of E. coli) | 1-2 days after ingestion of lactulose
  microbiota sequencing, analysis of E. coli

SECONDARY OUTCOMES:
Influence of lactulose intake on metabolic profiles within the fecal ecoystem (metabolomics analysis) | 1-2 days after ingestion of lactulose
  metabolomics analysis
Correlation of gut microbiota composition and H2-peak (H2-measurements) | within 3 hours after lactulose ingestion
  H2-measurements
Correlation of gut microbiota composition and symptoms (standardized record of symptoms) | within 3 hours after lactulose ingestion
  standardized record of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, MD, Principal Investigator — University of Zurich; Gerhard Rogler, MD PhD, Study Chair — University of Zurich
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Wotzka SY, Kreuzer M, Maier L, Zund M, Schlumberger M, Nguyen B, Fox M, Pohl D, Heinrich H, Rogler G, Biedermann L, Scharl M, Sunagawa S, Hardt WD, Misselwitz B. Microbiota stability in healthy individuals after single-dose lactulose challenge-A randomized controlled study. PLoS One. 2018 Oct 25;13(10):e0206214. doi: 10.1371/journal.pone.0206214. eCollection 2018. PMID 30359438